CLINICAL TRIAL: NCT03722953
Title: The Role of Shear Stress in the Cerebrovascular Response to Acute Exercise
Brief Title: Cerebrovascular Response to Acute Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-0783; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison); Protocol Version 10/23/2018 (Other: UW Madison)
Record Dates: First submitted 2018-10-15; First posted 2018-10-29 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2022-06

CONDITIONS: Healthy; Physical Activity
Keywords: Exercise; Treadmill; Vascular Function; Intensity
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic Exercise (Other): Control: Cerebrovascular function and peripheral vascular function will be measured.
  Aerobic Exercise: Across four separate visits, participants will perform light intensity exercise, light intensity exercise plus an additional task, vigorous intensity exercise and vigorous intensity exercise to match the energy expenditure of light intensity exercise visit.
  Interventions: Other: Control; Other: Aerobic Exercise

INTERVENTIONS:
Other: Control — 1. Ultrasound
  2. Blood Pressure
  3. Heart Rate
  4. Oxygen Saturation
Other: Aerobic Exercise — 1. Ultrasound
  2. Blood Pressure
  3. Heart Rate
  4. Oxygen Saturation

SUMMARY:
Cerebrovascular function and peripheral vascular function will be measured in healthy young adults, before and after acute bouts of aerobic exercise at various intensities.

DETAILED DESCRIPTION:
Acute bouts of aerobic exercise have been shown to enhance vascular reactivity of the peripheral circulation; however, the effects of a single exercise session on the cerebral circulation are unknown. This study will measure cerebrovascular function and peripheral vascular function before and after aerobic exercise at high and low intensities.

The research aims are:

1. To determine if a single bout of aerobic exercise acutely enhances cerebrovascular function
2. To determine the effect of aerobic exercise intensity and dose on cerebrovascular function in healthy adults.
3. To determine if the acute exercise-induced changes in cerebrovascular function are associated with acute exercise-induced changes in peripheral vascular function in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-40 years old
* BMI < 30 kg/m2
* Recreationally active
* Experience running on a treadmill

Exclusion Criteria:

* Current smoker
* History or evidence of: hepatic disease, renal disease, hematological disease, cardiovascular disease, stroke/neurovascular disease, diabetes
* Taking blood pressure medication
* History of depression or other mood related disorders
* Part of a vulnerable population (e.g. pregnant women, prisoner, individuals lacking capacity to consent, etc.)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular function | Change in cerebrovascular function: measurements occur at baseline and 90 minutes post aerobic exercise to quantify magnitude of change.
  Utilize ultrasound to measure a change in blood flow velocity in response to a breathing test
Peripheral vascular function | Change in peripheral vascular function: measurements occur at baseline and 60 minutes post aerobic exercise to quantify magnitude of change.
  Utilize ultrasound to measure a change in brachial artery diameter in response to reactive hyperemia

CONTACTS AND LOCATIONS:
Locations (1):
- Gymnasium-Natatorium, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes JN, Schmidt JE, Nicholson WT, Joyner MJ. Cyclooxygenase inhibition abolishes age-related differences in cerebral vasodilator responses to hypercapnia. J Appl Physiol (1985). 2012 Jun;112(11):1884-90. doi: 10.1152/japplphysiol.01270.2011. Epub 2012 Mar 22. PMID 22442028
- [Background] Richiardi J, Monsch AU, Haas T, Barkhof F, Van de Ville D, Radu EW, Kressig RW, Haller S. Altered cerebrovascular reactivity velocity in mild cognitive impairment and Alzheimer's disease. Neurobiol Aging. 2015 Jan;36(1):33-41. doi: 10.1016/j.neurobiolaging.2014.07.020. Epub 2014 Jul 24. PMID 25146454
- [Background] Sam K, Crawley AP, Conklin J, Poublanc J, Sobczyk O, Mandell DM, Venkatraghavan L, Duffin J, Fisher JA, Black SE, Mikulis DJ. Development of White Matter Hyperintensity Is Preceded by Reduced Cerebrovascular Reactivity. Ann Neurol. 2016 Aug;80(2):277-85. doi: 10.1002/ana.24712. PMID 27352039
- [Background] Shin HK, Jones PB, Garcia-Alloza M, Borrelli L, Greenberg SM, Bacskai BJ, Frosch MP, Hyman BT, Moskowitz MA, Ayata C. Age-dependent cerebrovascular dysfunction in a transgenic mouse model of cerebral amyloid angiopathy. Brain. 2007 Sep;130(Pt 9):2310-9. doi: 10.1093/brain/awm156. Epub 2007 Jul 16. PMID 17638859
- [Background] Barnes JN, Taylor JL, Kluck BN, Johnson CP, Joyner MJ. Cerebrovascular reactivity is associated with maximal aerobic capacity in healthy older adults. J Appl Physiol (1985). 2013 May 15;114(10):1383-7. doi: 10.1152/japplphysiol.01258.2012. Epub 2013 Mar 7. PMID 23471946
- [Background] Tarumi T, Zhang R. Cerebral hemodynamics of the aging brain: risk of Alzheimer disease and benefit of aerobic exercise. Front Physiol. 2014 Jan 21;5:6. doi: 10.3389/fphys.2014.00006. eCollection 2014. PMID 24478719
- [Background] Mitchell GF. Effects of central arterial aging on the structure and function of the peripheral vasculature: implications for end-organ damage. J Appl Physiol (1985). 2008 Nov;105(5):1652-60. doi: 10.1152/japplphysiol.90549.2008. Epub 2008 Sep 4. PMID 18772322
- [Background] Ranjan V, Xiao Z, Diamond SL. Constitutive NOS expression in cultured endothelial cells is elevated by fluid shear stress. Am J Physiol. 1995 Aug;269(2 Pt 2):H550-5. doi: 10.1152/ajpheart.1995.269.2.H550. PMID 7544542
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Endres M, Gertz K, Lindauer U, Katchanov J, Schultze J, Schrock H, Nickenig G, Kuschinsky W, Dirnagl U, Laufs U. Mechanisms of stroke protection by physical activity. Ann Neurol. 2003 Nov;54(5):582-90. doi: 10.1002/ana.10722. PMID 14595647
- [Background] Tinken TM, Thijssen DH, Hopkins N, Black MA, Dawson EA, Minson CT, Newcomer SC, Laughlin MH, Cable NT, Green DJ. Impact of shear rate modulation on vascular function in humans. Hypertension. 2009 Aug;54(2):278-85. doi: 10.1161/HYPERTENSIONAHA.109.134361. Epub 2009 Jun 22. PMID 19546374
- [Background] Dawson EA, Green DJ, Cable NT, Thijssen DH. Effects of acute exercise on flow-mediated dilatation in healthy humans. J Appl Physiol (1985). 2013 Dec;115(11):1589-98. doi: 10.1152/japplphysiol.00450.2013. Epub 2013 Sep 12. PMID 24030665
- [Background] Iadecola C, Zhang F. Nitric oxide-dependent and -independent components of cerebrovasodilation elicited by hypercapnia. Am J Physiol. 1994 Feb;266(2 Pt 2):R546-52. doi: 10.1152/ajpregu.1994.266.2.R546. PMID 7511352
- [Background] Molina C, Sabin JA, Montaner J, Rovira A, Abilleira S, Codina A. Impaired cerebrovascular reactivity as a risk marker for first-ever lacunar infarction: A case-control study. Stroke. 1999 Nov;30(11):2296-301. doi: 10.1161/01.str.30.11.2296. PMID 10548661
- [Background] Buratti L, Viticchi G, Falsetti L, Balucani C, Altamura C, Petrelli C, Provinciali L, Vernieri F, Silvestrini M. Thresholds of impaired cerebral hemodynamics that predict short-term cognitive decline in asymptomatic carotid stenosis. J Cereb Blood Flow Metab. 2016 Oct;36(10):1804-1812. doi: 10.1177/0271678X15613526. Epub 2015 Oct 27. PMID 26661219
- [Background] Moraine JJ, Lamotte M, Berre J, Niset G, Leduc A, Naeije R. Relationship of middle cerebral artery blood flow velocity to intensity during dynamic exercise in normal subjects. Eur J Appl Physiol Occup Physiol. 1993;67(1):35-8. doi: 10.1007/BF00377701. PMID 8375362
- [Background] Ide K, Secher NH. Cerebral blood flow and metabolism during exercise. Prog Neurobiol. 2000 Jul;61(4):397-414. doi: 10.1016/s0301-0082(99)00057-x. PMID 10727781
- [Background] Barnes JN, Harvey RE, Miller KB, Jayachandran M, Malterer KR, Lahr BD, Bailey KR, Joyner MJ, Miller VM. Cerebrovascular Reactivity and Vascular Activation in Postmenopausal Women With Histories of Preeclampsia. Hypertension. 2018 Jan;71(1):110-117. doi: 10.1161/HYPERTENSIONAHA.117.10248. Epub 2017 Nov 20. PMID 29158356
- [Background] Miller KB, Howery AJ, Harvey RE, Eldridge MW, Barnes JN. Cerebrovascular Reactivity and Central Arterial Stiffness in Habitually Exercising Healthy Adults. Front Physiol. 2018 Aug 17;9:1096. doi: 10.3389/fphys.2018.01096. eCollection 2018. PMID 30174609
- [Background] Morrell MJ, Harty HR, Adams L, Guz A. Changes in total pulmonary resistance and PCO2 between wakefulness and sleep in normal human subjects. J Appl Physiol (1985). 1995 Apr;78(4):1339-49. doi: 10.1152/jappl.1995.78.4.1339. PMID 7615441
- [Background] Meza S, Mendez M, Ostrowski M, Younes M. Susceptibility to periodic breathing with assisted ventilation during sleep in normal subjects. J Appl Physiol (1985). 1998 Nov;85(5):1929-40. doi: 10.1152/jappl.1998.85.5.1929. PMID 9804601
- [Background] Barnes JN, Nualnim N, Dhindsa M, Renzi CP, Tanaka H. Macro- and microvascular function in habitually exercising systemic lupus erythematosus patients. Scand J Rheumatol. 2014;43(3):209-16. doi: 10.3109/03009742.2013.846408. Epub 2014 Jan 7. PMID 24392783
- [Background] Dhindsa M, Sommerlad SM, DeVan AE, Barnes JN, Sugawara J, Ley O, Tanaka H. Interrelationships among noninvasive measures of postischemic macro- and microvascular reactivity. J Appl Physiol (1985). 2008 Aug;105(2):427-32. doi: 10.1152/japplphysiol.90431.2008. Epub 2008 May 15. PMID 18483158
- [Background] Ogoh S, Sorensen H, Hirasawa A, Sasaki H, Washio T, Hashimoto T, Bailey DM, Secher NH. Dynamic cerebral autoregulation is unrelated to decrease in external carotid artery blood flow during acute hypotension in healthy young men. Exp Physiol. 2016 Aug 1;101(8):1040-9. doi: 10.1113/EP085772. Epub 2016 Jun 21. PMID 27228963
- [Background] Tanaka H, Shimizu S, Ohmori F, Muraoka Y, Kumagai M, Yoshizawa M, Kagaya A. Increases in blood flow and shear stress to nonworking limbs during incremental exercise. Med Sci Sports Exerc. 2006 Jan;38(1):81-5. doi: 10.1249/01.mss.0000191166.81789.de. PMID 16394957